CLINICAL TRIAL: NCT04031677
Title: A Randomized Phase III Study of Neoadjuvant Chemotherapy Followed by Surgery Versus Surgery Alone for Patients With High Risk RetroPeritoneal Sarcoma (RPS)
Brief Title: Surgery With or Without Neoadjuvant Chemotherapy in High Risk RetroPeritoneal Sarcoma
Acronym: STRASS2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Canadian Cancer Trials Group (Network); ECOG-ACRIN Cancer Research Group (Network); Anticancer Fund, Belgium (Other); Australia and New Zealand Sarcoma Association (Other); Japan Clinical Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 1809-STBSG; EA7211 (Other: ECOG-ACRIN Cancer Research Group); SR.7 (Other: Canadian Cancer Trials Group); ASSG45 (Other: Australia and New Zealand Sarcoma Association); JCOG2214INT (Other: Japan Clinical Oncology Group)
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Retroperitoneal Sarcoma; Liposarcoma; Leiomyosarcoma
MeSH Terms: conditions — Liposarcoma; Leiomyosarcoma | interventions — Surgical Procedures, Operative; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard arm (Other): Surgery alone
  Interventions: Procedure: Surgery
- Experimental arm (Experimental): Preoperative chemotherapy and surgery
  Interventions: Drug: Preoperative chemotherapy

INTERVENTIONS:
Procedure: Surgery — Large en-bloc curative-intent surgery
  Arms: Standard arm
Drug: Preoperative chemotherapy — * High grade LPS: ADM 75 mg/m2 (or the equivalent EpiADM 120 mg/m2) + ifosfamide 9 g/m2 Q3 weeks
  * LMS: ADM 75 mg/m2 + DTIC 1g/m2 Q3 weeks
  Note: the recommended dose of Doxorubicin (or Epirubicin) can be modified according to national/institutional guidelines, given that the minimal threshold must be Doxorubicin 60 mg/m2 per cycle (or the equivalent Epirubicin 95 mg/m2 per cycle); the recommended dose of Ifosfamide can be modified according to national/institutional guidelines, given that the minimal threshold must be 7.5 g/m2 per cycle; the recommended dose of Dacarbazine can be modified according to national/institutional guidelines, given that the minimal threshold must be 900 mg/m2 per cycle. The schedule of administration of above chemotherapies can be modified according to national/institutional guidelines provided that the minimal threshold of doses, and the treatment periods with chemotherapies remain the same.
  Other Names: neoadjuvant chemotherapy
  Arms: Experimental arm

SUMMARY:
This is a multicenter, randomized, open label phase lll trial to assess whether preoperative chemotherapy, as an adjunct to curative-intent surgery, improves the prognosis of high risk DDLPS (dedifferentiated Liposarcoma) and LMS (Leiomyosarcoma) patients as measured by disease free survival.

After confirmation of eligibility criteria, patients will be randomized to either the standard arm or experimental arm.

DETAILED DESCRIPTION:
Standard arm:

* Large en-bloc curative-intent surgery within 4 weeks following randomization- Experimental arm

Experimental arm:

* 3 cycles of neoadjuvant chemotherapy starting within 2 weeks following randomization:

  * High grade LPS: ADM (doxorubicin) 75 mg/m2 (or the equivalent EpiADM 120 mg/m2) + ifosfamide 9 g/m3 Q3 weeks.
  * LMS: ADM 75 mg/m2 + DTIC (dacarbazine) 1 g/m2 Q3 weeks
* re-assessment of operability
* curative-intent surgery within 3-6 weeks of last cycle of chemotherapy

ELIGIBILITY:
1. STRASS 2

   Inclusion Criteria:
   * Histologically proven primary high risk leiomyosarcoma (LMS) or Liposarcoma (LPS) of retroperitoneal space or infra-peritoneal spaces of pelvis.
   * LMS:

     * Any grade LMS can be included
     * Minimum size of LMS tumor should be 5 cm
   * LPS:

     * Diagnosis should be confirmed based on MDM2 (Mouse double minute 2 homolog) and CDK4 (Cyclin-dependent kinase 4) expression on IHC (immunohistochemistry), while proof of MDM2 amplification is highly recommended.
     * All grade 3 DDLPS can be included.
     * DDLPS with confirmed grade 2 on biopsy can be included when:

       * The grade 2 DDLPS has an FNCLCC score=5 (Fédération Nationale des Centres de Lutte Contre Le Cancer), and clear necrosis on imaging (whether or not present on the biopsy).
       * The tumors carry a high risk gene profile as determined by the Complexity INdex in SARComas (CINSARC-high)
     * Unifocal tumour
     * Resectable tumour: resectability is based on pre-operative imaging (CT-abdomen, potentially also with MRI) and has to be defined by the local treating sarcoma team. A patient is not considered resectable when the expectation is that only an R2 resection is feasible.
     * Criteria for non-resectability are:
     * Involvement of the superior mesenteric artery, aorta, coeliac trunk and/or portal vein
     * Involvement of bone
     * Growth into the spinal canal
     * Progression of retro-hepatic inferior vena cava leiomyosarcoma towards the right atrium
     * Infiltration of multiple major organs like liver, pancreas and or major vessels
     * Patient must have radiologically measurable disease (RECIST 1.1), as confirmed by imaging. CT thorax abdomen pelvis with IV contrast is the preferred imaging modality. In case of any contra-indications (medical or regulatory), it is allowed to perform a non-contrast CT thorax + MRI abdomen & pelvis
     * Collection of tumour tissue for central pathology review is mandatory.
     * For patients with LMS: if there is not enough tissue for assessing the grading, this is acceptable.
     * If tumour tissue is not available for the central pathology review, patient will not be eligible.
     * If the biopsy was not done or the FFPE of the biopsy not available but at least 10 unstained slides or one pathological block are available for the central review, that will be considered as acceptable.
     * For the biopsy if fine needle aspiration (FNA) is performed instead of core needle biopsy (CNB) recommended by the standard guidelines, please contact the EORTC medical monitors for further evaluation.
     * Collection of tumour tissue and blood samples for translational research is mandatory.
     * In case there is not enough tissue for TR, a new biopsy is not required and if the patient fulfils all other eligibility criteria, he/she will be eligible.
     * If the blood samples are not collected, patient will not be eligible.
     * If the patient refuses the collection of biomaterial for TR, patient will not be eligible even if he/she fulfils all other eligibility criteria
     * ≥ 18 years old (no upper age limit)
     * WHO performance status ≤ 2
     * Adequate haematological and organ function
     * American Society of Anaesthesiologist (ASA) score < 3
     * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 3 days prior to randomization.

   Note: a woman is considered of childbearing potential, i.e., fertile, if she is following menarche. She remains of childbearing potential until she becomes post-menopausal or permanently sterile.Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 consecutive months without menses, a single FSH measurement is insufficient.
   * WOCBP in both arms should use highly effective birth control measures, during the study treatment period and for at least 6 months after the last dose of chemotherapy or date of surgery (except for women receiving chemotherapy with ifosfamide who should continue contraception until 1 year after last day of treatment). A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.
   * For men in the experimental arm: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm.
   * Female subjects who are breast feeding should discontinue nursing prior to the first day of study treatment and until 6months after the last study treatment.
   * Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

   Exclusion criteria:
   * Sarcoma originating from bone structure, abdominal or gynecological viscera
   * Extension through the sciatic notch or across the diaphragm
   * Metastatic disease
   * Any previous surgery (excluding diagnostic biopsy), radiotherapy or systemic therapy for the present tumour
   * Hypersensitivity to doxorubicin, ifosfamide, dacarbazine or to any of their metabolites or to any of their excipients
   * Congestive heart failure
   * Angina pectoris
   * Myocardial infarction within 1 year before randomization
   * Uncontrolled arterial hypertension defined as blood pressure ≥ 150/100 mm Hg despite optimal medical therapy.

   Note: in case of high blood pressure: 1) initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry; 2) blood pressure must be re-assessed on two occasions that are separated by a minimum of 1 hour. The mean SBP / DBP values from each blood pressure assessment must be ≤ 150/90mmHg in order for a patient to be eligible for the study.
   * Uncontrolled cardiac arrhythmia
   * Previous treatment with maximum cumulative doses (450mg/m² Doxorubicin or equivalent 900mg/m² Epirubicin) of doxorubicin, daunorubicin, epirubicin, idarubicin, and/or other anthracyclines and anthracenediones
   * Active and uncontrolled infections
   * Vaccination with live vaccines within 30 days prior to study entry
   * Inflammation of the urinary bladder (interstitial cystitis) and/or obstructions of the urine flow.
   * Other invasive malignancy within 5 years, with the exception of adequately treated non-melanoma skin cancer, localized cervical cancer, localized and Gleason ≤ 6prostate cancer.
   * Uncontrolled severe illness, infection, medical condition (including uncontrolled diabetes), other than the primary LPS or LMS of the retroperitoneum.
   * Female patients who are pregnant or breastfeeding or female and male patients of reproductive potential who are not willing to employ effective birth control method.
   * Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial
   * Known contraindication to imaging tracer and to MRI
2. Selection criteria for STREXIT 2

   * Patients with histologically proven primary resectable localized high-risk DDLPS or LMS of retroperitoneal space or infra-peritoneal spaces of pelvis (as described in the inclusion criteria of STRASS 2) and amenable to receive chemotherapy but for whom the list of eligibility criteria for the study is too restrictive (tumour grading not available, inadequate organ function, concomitant diseases)
   * Patients who meet all eligibility criteria of STRASS 2 but do not consent to randomization or are not enrolled for any other reason.
   * Patients enrolled in a Registry collecting data on primary RPS patients in the centres participating in STRASS 2 (e.g., RESAR) and who satisfy the above criteria.
3. Selection criteria for preferences for neoadjuvant chemotherapy in STRASS 2 substudy

All patients recruited to STRASS 2 in participating centres (Australia +/- international sites) that are able to read, comprehend and write in English at a sufficient level to complete study materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2027-04-21 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 7 years from first patient in
  Disease free survival will be measured from the date of randomization (as reference) to the date of recurrence or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 8 years from first patient in
  OS will be measured from the date of randomization to the date of death, whatever the cause. Alive patients will be censored at the date of last follow-up.
Recurrence free survival | 8 years from first patient in
  Recurrence free survival will be measured in patients who were successfully operated (R0/R1 resection) from the date of surgery (as reference) to the date of recurrence (local or distant) or death, whichever occurs first. Patients without one of these events will be censored at the date of last follow-up.
Distant metastases free survival | 8 years from first patient in
  Distant metastases free survival will be from the date of randomization (as reference) to the date of distant metastases or death (whatever the cause), whichever occurs first. Patients without any of these events will be censored at the date of last follow-up.
Cumulative incidence of local recurrences | 8 years from first patient in
  Cumulative incidence of local recurrences will be measured from the date of randomization (as reference) to the date of local recurrence.
Cumulative incidence of distant metastases | 8 years from first patient in
  Cumulative incidence of distant metastases will be measured from the date of randomization to the date of occurrence of distant metastases.
Radiological response to neoadjuvant chemotherapy according to RECIST | 8 years from first patient in
  For patients receiving neo-adjuvant chemotherapy, the radiological response will be assessed using RECIST 1.1 by comparison of the baseline and preoperative imaging.
Radiological response to neoadjuvant chemotherapy according to CHOI | 8 years from first patient in
  For patients receiving neo-adjuvant chemotherapy, the radiological response will be also assessed using Choi criteria by comparison of the baseline and preoperative imaging.
Pathological response | 8 years from first patient in
  Response evaluation will be done according to the EORTC response score.
Safety and toxicity of neoadjuvant chemotherapy | 8 years from first patient in
  Safety and toxicity of neoadjuvant chemotherapy will be evaluated and graded using CTCAE V5.0.
Perioperative complications | 8 years from first patient in
  Perioperative complications will be evaluated with the Dindo scale for the events related to the surgery and CTCAE V5.0 will be used for all other events.
Late complications | 8 years from first patient in
  Late complications (after the 60th day following the surgery) will be evaluated and graded according to the CTCAE version 5.0.
Health-Related Quality of life (EORTC QLQ-C30 + Item list from QLQ-STO22) | 8 years from first patient in
  Health-Related Quality of life assessment will be based on the EORTC QLQ C30 questionnaire version 3.0, with additional questions from the QLQ-STO22 module.
Health utility, calculated from the collected patient-reported HRQoL data and patient demographics economics. | 8 years from first patient in
  he EORTC QLQ C30 data will be mapped to health utility values using an established indirect mapping approach.

CONTACTS AND LOCATIONS:
Locations (149):
- United States (91):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC Irvine Health/Chao Family Comprehensive Ca Ctr, Orange, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guiford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Ctr at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois at Chicago MBCCOP, Chicago, Illinois
  - Indiana Univ/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Ctr, Westwood, Kansas
  - James Graham Brown Ca Ctr at Univ of Louisville, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of The Lake Hospital, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Johns Hopkins Univ/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center-West County, Creve Coeur, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center-South Country, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Bellevue, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Med Ctr/Dartmouth Cancer Ctr, Lebanon, New Hampshire
  - HMH-Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Issac Perlmutter Ca Ctr at NYU Langone, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Cancer Center at Hanover Medical Park, Mechanicsville, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth Univ/Massey Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center, Minocqua, Wisconsin
  - Marshfield Medical Center, Rice Lake, Wisconsin
  - Marshfield Med Ctr-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center, Weston, Wisconsin
- Australia (3):
  - Princess Alexandra Hospital - University Of Queensland, Woolloongabba, Queensland
  - Peter Maccallum Cancer Institute, Melbourne, Victoria
  - Chris O'Brian Life House - Chris O'Brien Lifehouse, Camperdown
- Canada (6):
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Center, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hopital Maisonneuve Rosemont, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Mount Sinai Hospital, Toronto
- Bank Of Cyprus Oncology Centre, Stróvolos, Cyprus
- Masaryk Memorial Cancer Institute, Brno, Czechia
- Denmark (2):
  - Herlev Hospital - University Copenhagen, Herlev, Copenhagen
  - Aarhus University Hospitals - Aarhus University Hospital-Skejby, Aarhus
- France (5):
  - Centre Leon Berard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie- Hopital de Paris, Paris
  - Hopitaux Universitaires de Strasbourg - Hautepierre, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Universitaetsmedizin Goettingen - Georg-August Universitaet, Goettigen, Lower Saxony
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - UniversitaetsMedizin Mannheim, Mannheim
- Italy (8):
  - Centro Di Riferimento Oncologico, Aviano
  - IRCCS - Fondazione Piemonte Inst di Candiolo, Candiolo
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola
  - IRCCS - Istituto Nazionale dei Tumori, Milan
  - Istituto Clinico Humanitas, Milan
  - Istituto Europeo di Oncologia, Milan
  - IRCCS - Istituto Oncologico Veneto, Padua
  - Policlinico Universitario Campus Bio-Medico- Oncology Center, Roma
- Japan (12):
  - Kyushu University Hospital, Higashiku, Fukuoka
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Aichi Cancer Center, Chikusa-ku, Nagoya
  - Nagoya University Hospital, Shōwaku, Nagoya
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - Okayama University Hospital, Kita-ku, Okayama-ken
  - Osaka International Cancer Institute, Chuo-ku, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Saitama Medical Center, Jichi Medical University, Saitama
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Leiden University Medical Centre, Leiden
  - Radboudumc - Radboud University Medical Center Nijmegen, Nijmegen
- Maria Sklodowska-Curie Memorial Cancer Centre - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw, Poland
- National Cancer Institute, Bratislava, Slovakia
- Spain (4):
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Catala d'Oncologia - ICO Badalona - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario San Carlos, Madrid
- United Kingdom (8):
  - University Hospitals Birmingham - Queen Elisabeth Medical Centre, Birmingham
  - NHS Greater Glasgow and Clyde - Beatson West of Scotland Cancer Centre - Gartnavel General Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - the Royal Marsden Hospital, London
  - Clatterbridge cancer center, Metropolitan Borough of Wirral
  - Newcastle Hospitals - Freeman Hospital, Northern Centre For Cancer Care, Newcastle
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Oxford University Hospitals NHS Trust - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No